CLINICAL TRIAL: NCT01902069
Title: The Gut-brain Axis in Food Reward and Alcohol Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1305012106; 5P50AA012870 (NIH)
Record Dates: First submitted 2013-07-15; First posted 2013-07-17 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Impulsivity; Alcohol Consumption
Keywords: sweet and fat preference
MeSH Terms: conditions — Impulsive Behavior; Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phosholean dietary supplement (Experimental): Subjects in the PhosphoLean group will receive two capsules of PhosphoLEAN orally daily (total of 55 mg of NOPE and 100 mg of EGCG), one capsule consumed 60 minutes prior to lunch and one capsule 60 minutes prior to dinner.
  Interventions: Dietary Supplement: Phospholean
- Placebo (rice flour) group (Placebo Comparator): The control (placebo) group will receive a placebo (identical in appearance, but containing 100 mg of rice flour per capsule), one capsule consumed 60 minutes prior to lunch and one capsule 60 minutes prior to dinner.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phospholean — Phospholean supplied by Cheminutra (White Bear Lake, MN). PhosphoLean® N-Oleoyl-PE + EGCG (NOPE + EGCG) is a proprietary phosphobioflavonic complex of N-oleoyl-phosphatidyl-ethanolamine (NOPE), which contains oleoyl ethanolamine (OEA) bound to phosphatidylethanolamine (PE), and epigallocatechin gallate (EGCG).
  PhosphoLean® 40P is a dietary ingredient under the Dietary Supplement Health and Education Act (DSHEA) regulations of the US FDA (1994).
  Arms: Phosholean dietary supplement
Dietary Supplement: Placebo — Placebo consists of rice flour
  Arms: Placebo (rice flour) group

SUMMARY:
The aims of this project are to:

1. Determine if 3-weeks dietary supplementation with NOPE-EGCG (PhosphoLEANtm, 85mg NOPE+50mg EGCG per capsule) versus a placebo will improve performance on impulsivity, go/no-go tasks and negative outcome learning in heavy drinkers.
2. Evaluate whether supplementation with NOPE-EGCG versus placebo results in reductions in alcohol consumption.
3. Preliminary data in the rodent model suggests that rats treated with OEA shift preference for lower fat test stimuli. In aim 3 we will Determine if 3-weeks of supplementation with PhosphoLEAN shifts fat preference towards lower fat test puddings.

DETAILED DESCRIPTION:
Similarities in striatocortical pathway dysfunction have been noted for alcoholism and obesity. In prior studies we have demonstrated an inverse relationship between body mass index and response in the dorsal striatum (DS) during consumption of a palatable milkshake[1]. We have also shown that the magnitude of the reduced response predicts weight gain, especially in individuals who carry a copy of the A1 allele of the taq1A polymorphism[1]. Since the A1 allele is associated with reduced striatal D2 receptors [2-7], this finding implicates the dopamine system in the reduced blood oxygen level dependent (BOLD) response. Our results also indicate that this reduced response is a consequence, rather than a cause of obesity, since gaining weight [8], but not risk for obesity [9] (by virtue of parental obesity), is associated with reduced DS response to palatable food. Taken together the results indicate that increased adiposity is associated with blunted DS response to palatable food that may reflect altered dopamine signaling. More recently we determined that reduced DS responses in overweight and obese subjects are associated with increased impulsivity measured with the BIS-11 and a go no/no-go task [10]. Heavy drinkers are also more likely to be impulsive [11]. In preliminary analyses of data on over 300 individuals assessed with the clinical core battery in the Center for the Translational Neuroscience of Alcoholism (CTNA), we found that higher scores on the BIS-11 and other measures of impulsivity were associated with greater alcohol consumption.

Related to these findings in humans, preliminary work in rodents shows that exogenous administration of N-Acylethanolamines, such as oleoylethanolamine (OEA) can normalize high-fat diet induced dopamine decreases in DS. Human testing of OEA supplementation is possible based on the availability of a dietary supplement containing the OEA precursor NOPE-EGCG ((PhosphoLEANtm, 85mg NOPE+50mg EGCG per capsule). PhosphoLEAN has been shown to enhance adherence to dietary advice in overweight healthy subjects [12-14]. We therefore propose a pilot study to test whether PhosphoLEAN will improve performance on impulsivity, go/no-go tasks and negative outcome learning. Specifically, we will recruit heavy drinkers because they are more likely to be impulsive [11]. Phospholean may improve negative reinforcement learning in this population. This may lead to reductions in drinking as well. We will also explore whether the supplement leads to reductions in alcohol consumption and preference for high fat foods.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting NIAAA heavy drinking criteria (for men defined as consuming 5 or more standard drinks on a drinking day and for women as consuming 4 or more standard drinks on a drinking day at least once per week for the prior 30 days, with an upper limit of 40 standard drinks per week). Half will be women. Right handed, English speaking, be a non-smoker (never smoked more than 2 cigarettes per month). Subjects will have a BMI between 18.5 and 35.

Exclusion Criteria:

* a) serious or unstable medical illness (e.g., cancer); b) past or current history of alcoholism or consistent drug use; c) current major psychiatric illness as defined by the DSM-IV criteria including eating disorders d) medications that affect alertness (e.g., barbiturates, benzodiazepines, chloral hydrate, haloperidol, lithium, carbamazepine, phenytoin, etc.); e) history of major head trauma with loss of consciousness; f) ongoing pregnancy; g) known taste or smell dysfunction; h) a diagnosis of diabetes; i) any known food allergy, certain food sensitivities (lactose); j) pregnant or nursing women. Daily drinkers and individuals meeting criteria for alcohol dependence will be excluded.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Fat and sweet preference | 21 days
  Subject will be asked to sample and rate fatty and sweet flavor stimuli (all made from commercially available ingredients).
Impulsivity | 21 days
  Various questionnaires and computer tasks addressing impulsivity.
Alcohol consumption | 21 days
  Interview addressing alcohol consumption

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Small, PhD, Principal Investigator — The John B. Pierce Laboratory
Locations (1):
- John B Pierce Laboratory, New Haven, Connecticut, United States